CLINICAL TRIAL: NCT06224946
Title: IMPACT OF THE SOLUBLE LIKE TYROSINE KINASE/PLACENTAL GROWTH FACTOR RATIO ON MEDICAL DECISION-MAKING AND ON MATERNAL AND NEONATAL OUTCOMES IN WOMEN SUSPECTED OF PREECLAMPSIA
Brief Title: IMPACT OF THE BIOLOGICAL RATIO ON MEDICAL DECISION MAKING IN WOMEN SUSPECTED OF PREECLAMPSIA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: CEROG 2022-OBS-0401
Record Dates: First submitted 2024-01-09; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Pre-Eclampsia
Keywords: Pre-Eclampsia; Placental Growth Factor; Soluble fms-like tyrosine Kinase; medical Care decision
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women under 37 weeks of gestation age: 217 women under 37 weeks of gestation age
  Interventions: Diagnostic Test: soluble fms-like tyrosine kinase (sFlt-1) / placental growth factor (PlGF) ratio
- women above 37 weeks of gestation age: 97 women above 37 weeks of gestation age
  Interventions: Diagnostic Test: soluble fms-like tyrosine kinase (sFlt-1) / placental growth factor (PlGF) ratio

INTERVENTIONS:
Diagnostic Test: soluble fms-like tyrosine kinase (sFlt-1) / placental growth factor (PlGF) ratio — the soluble fms-like tyrosine kinase (sFlt-1) / placental growth factor (PlGF) ratio for pre-eclampsia diagnostic

SUMMARY:
Previous studies demonstrated that Placental Growth Factor (PIGF) and Vascular Endothelial Growth Factor (VEGF) produced by trophoblast cells decreases during Preeclampsia, whereas soluble fms-like tyrosine kinase-1 (sFlt-1), an antiangiogenic factor, increases. The ratio sFlt-1/PlGF has a higher positive predictive value than the isolated measurement. A ratio under 38 exclude risk of imminent preeclampsia and allows to outpatient follow-up with a negative predictive value of 99.3%. A ratio equal or higher than 38 permits to direct high-risk patients towards hospitalization with a positive predictive value of 36.7% of preeclampsia at 4 weeks. These findings suggest that the ratio can be used to select more appropriately women needing hospitalization for suspected preeclampsia.

This is a single-center prospective and observational study conducted from the 1rst of October 2019 to the 27th of January 2021, including pregnant women suspected of preeclampsia, above 24 weeks of gestation. Values were measured using the Elecsys sFlt-1/PlGF immunoassay ratio. The aim of the study is to observe the clinical decision regarding hospitalization, intensive patient monitoring, corticosteroid administration, and labor induction before and after knowing the ratio value

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients over 24 weeks of amenorrhea
* aged 18 and over
* with suspicion of preeclampsia defined by the appearance of pregnancy-induced hypertension (≥ 140 in systolic and/or 90 mmHg in diastolic pressure over 2 measurements at 4 hours intervals) OR proteinuria (≥ 0.3 g per 24 hours).
* who systematically gave oral consent after submitting the information sheet

Exclusion Criteria:

* pregnant women with both hypertension and proteinuria because they already have a confirmed diagnosis of preeclampsia.
* receiving antihypertensive treatment before pregnancy
* or refusing to participate in the study The sFlt-1/PlGF ratio was measured only when clinically indicated as per the investigator's judgment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 314 patients were included: 217 women under 37 weeks of gestation age and 97 women above this age.
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
The soluble fms-like tyrosine kinase (sFlt-1) / placental growth factor (PlGF) ratio | day 1
  Evaluate the impact of the soluble fms-like tyrosine kinase (sFlt-1) / placental growth factor (PlGF) ratio on medical decision-making in women with suspected preeclampsia in routine medical care.

CONTACTS AND LOCATIONS:
Overall Officials: BARJAT Tiphaine, MD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No